CLINICAL TRIAL: NCT07346976
Title: Investigation Into the Dynamic Variations of End-Tidal Carbon Monoxide Concentration (ETCOc) in Neonates Utilizing Non-Dispersive Infrared Spectroscopy and Its Implications for Jaundice Management.
Acronym: ETCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KY-2025-182
Record Dates: First submitted 2025-12-03; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-06

CONDITIONS: Neonatal Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- term neonates (Experimental): The non-dispersive infrared spectroscopy technique was employed to measure the end-tidal carbon monoxide (ETCOc) levels in newborns at intervals of 12, 24, 48, and 72 hours post-birth.
  Interventions: Device: Erythrocyte Life Span Tester

INTERVENTIONS:
Device: Erythrocyte Life Span Tester — The non-dispersive infrared spectroscopy technique was employed to measure the end-tidal carbon monoxide (ETCOc) levels in newborns at intervals of 12, 24, 48, and 72 hours post-birth.

SUMMARY:
The objective of this study is to ascertain the diagnostic threshold of end-tidal carbon monoxide (ETCOc, adjusted for ambient CO levels) within the first three days postpartum, stratified by neonatal age at birth. Additionally, the study aims to evaluate the concordance of the risk range of ETCOc, as measured by non-dispersive infrared spectroscopy, with existing literature, and to assess the reliability of this technology in the management of neonatal hyperbilirubinemia.

ELIGIBILITY:
Inclusion Criteria:

1. Newborns with gestational age of ≥ 37 weeks and birth weight of ≥ 2.5 kg;
2. Newborns delivered by either vaginal delivery or cesarean section and with hospital stay of ≥ 3 days.

Exclusion Criteria:

1. History of second-hand smoke exposure within 24 hours
2. Parents smoke or are exposed to second-hand smoke.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The ETCOc values of newborns were measured, and the optimal ETCOc threshold values between different time points of the TSB group were obtained. | The non-dispersive infrared spectroscopy technique was used to detect ETCOc in newborns at 12 hours, 24 hours, 48 hours and 72 hours after birth (the ETCOc detection should be completed within 4 hours at each time point)
  Establish an ETCOc diagnostic threshold for assessing the risk of hyperbilirubinemia in the early postnatal period based on the infant's age at birth. Determine the reliability and repeatability of ETCOc detection using non-dispersive infrared spectroscopy technology.Compare the concentrations of ETCOc between different groups and employ the ROC curve method to ascertain the optimal cut-off values of ETCOc at various time points across the TSB groups.
The ETCOc values of newborns | 12 hours, 24 hours, 48 hours and 72 hours after the birth of the newborn
  The ETCOc values of newborns were measured, and the optimal ETCOc threshold values between different time points of the TSB group were obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- 4th Affiliated Hospital, School of Medicine, Zhejiang University, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No